CLINICAL TRIAL: NCT01357148
Title: Sitagliptin Phosphate/Metformin HCl (JANUMET®) Post Marketing Surveillance Protocol
Brief Title: A Post Marketing Safety Study of Sitagliptin Phosphate/Metformin Hydrochloride (JANUMET®) (MK-0431A-235)
Status: Terminated | Type: Observational
Why Stopped: Completion of MK-0431A-235 was rendered unnecessary, as the local oversight authority accepted in its stead the results of another study [MK-0431-234].
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0431A-235
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants treated with sitagliptin phosphate/metformin HCl
  Interventions: Drug: Sitagliptin Phosphate/Metformin HCl (JANUMET®)

INTERVENTIONS:
Drug: Sitagliptin Phosphate/Metformin HCl (JANUMET®) — Participants prescribed Sitagliptin Phosphate/Metformin HCl (JANUMET®) in routine clinical practice.

SUMMARY:
The primary objective of this study is to obtain safety information on the use of sitagliptin phosphate/metformin hydrochloride (HCl) (JANUMET®) from endocrinologists, diabetologists, internists, and general practitioners.

ELIGIBILITY:
Inclusion Criteria:

* Must be taking sitagliptin phosphate/metformin HCl (JANUMET®) for the treatment of type 2 diabetes mellitus
* Treating physician must agree to provide information regarding the participant's treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with type 2 diabetes mellitus who are treated with sitagliptin phosphate/metformin HCl as per the standard of care in a physician's practice
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a postmarketing, safety study of participants with Type 2 diabetes mellitus prescribed sitagliptin phosphate/metformin HCL (JANUMET®) in clinical practices in the Philippines from January 2009 to May 2010.
Groups:
- Sitagliptin Phosphate/Metformin HCl: Participants prescribed sitagliptin phosphate/metformin HCl in routine clinical practice.
Period: Overall Study
Arm/Group | Sitagliptin Phosphate/Metformin HCl
Started | 143
Completed | 143
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sitagliptin Phosphate/Metformin HCl
Number analyzed (Participants) | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13.2)
Sex/Gender, Customized [Number; unit: participants]
  Female | 74
  Male | 66
  Unspecified | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Time Frame: Up to approximately 28 months
Measure: Number; unit: participants
Arm/Group | Sitagliptin Phosphate/Metformin HCl
Number analyzed (Participants) | 143
participants | 6

2. Primary Outcome: Age of Participants Prescribed Sitagliptin Phosphate/Metformin HCl
Time Frame: Up to approximately 28 months
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Sitagliptin Phosphate/Metformin HCl
Number analyzed (Participants) | 143
years | 51 (13.2)

3. Primary Outcome: Number of Participants With Concomitant Conditions
Time Frame: Up to approximately 28 months
Measure: Number; unit: participants
Arm/Group | Sitagliptin Phosphate/Metformin HCl
Number analyzed (Participants) | 143
participants | 100

4. Primary Outcome: Number of Participants Taking Concomitant Medications
Time Frame: Up to approximately 28 months
Measure: Number; unit: participants
Arm/Group | Sitagliptin Phosphate/Metformin HCl
Number analyzed (Participants) | 143
participants | 86

ADVERSE EVENTS:
Time Frame: Up to approximately 28 months
Arm/Group | Sitagliptin Phosphate/Metformin HCl
Serious Adverse Events (participants affected / at risk) | 0/143
Other Adverse Events (participants affected / at risk) | 0/143

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No